CLINICAL TRIAL: NCT00749996
Title: Herniectomy vs. Herniectomy With a Spinal Stabilization System for the Treatment of Complex Disc Disease
Brief Title: Herniectomy Versus Herniectomy With a Spinal Stabilization System for the Treatment of Complex Disc Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAM™ Study
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Sciatica; Back Pain
MeSH Terms: conditions — Sciatica; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational group (Experimental): Single level herniectomy followed by placement of the DIAM™ Spinal Stabilization System
  Interventions: Device: DIAM™ Spinal Stabilization System
- Control group (Active Comparator): Single level herniectomy
  Interventions: Procedure: Herniectomy

INTERVENTIONS:
Device: DIAM™ Spinal Stabilization System — The DIAM™ Spinal Stabilization System is a spacer that is inserted between adjoining spinous processes after doing a standard herniectomy procedure using a posterior surgical approach.
  Arms: Investigational group
Procedure: Herniectomy — Herniectomy is defined as the "removal of the extruded/protruded/sequestrated disc material". This is done by probing the annulus and disc space and removing all mobile disc fragments.
  Arms: Control group

SUMMARY:
The study aims at assessing the short and long-term effectiveness and patient perception of benefit with the use of a DIAM™ Spinal Stabilization System in the treatment of complex disc disease at a single level from L2 to L5.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized, controlled trial. Patients will be randomized in 2 groups:

Investigational group: a single level herniectomy procedure, followed by placement of the DIAMTM Spinal Stabilization System; Control group: a single level herniectomy procedure; After surgery, patients will be followed for a 2 years period with required follow up visits at 6 weeks, 3 months, 6 months, 1 year, 2 years and 4 years (optional visit).

ELIGIBILITY:
Inclusion Criteria:

* Has a history of sciatica (radicular pain) for at least 6 weeks, but not more than 1 year secondary to one symptomatic lumbar disc herniation at the levels L2-L5 as confirmed by patient history and clinical evaluation, and without major neurological impairment (i.e. not less than M 3/5; Medical Research Council Classification);
* Has a history of continuous low back pain for no more than 1 year secondary to lumbar degenerative disc disease (intermittent back pain may occur for more than a year);
* Has pre-treatment back pain score greater than or equal to 3, concomitant with leg pain score greater than or equal to 6. Leg pain score must be greater than back pain score (pain intensity score measured on a 10 cm VAS scale);
* Has one symptomatic disc herniation: protrusion, extrusion or sequestration (Milette & Fardon, 2001) as confirmed by MRI at the target level;
* Evidence of disc degeneration ≤ Grade IV at the target and adjacent levels as confirmed by MRI (Pfirrmann, 2001);
* Has an Oswestry Disability Index (ODI) score ≥ 34%;
* Has been treated non-operatively (e.g. bed rest, physical therapy, medications, TENS, manipulation, hydrotherapy, acupressure/acupuncture, massage, bracing and/or spinal injections) for at least 6 continuous weeks unless strong clinical grounds for expediting surgery;
* Patient male or female, age 20-60 years inclusive and is skeletally mature;
* Is willing and able to comply with the study plan and able to provide an informed consent;

Exclusion Criteria:

* Has a primary diagnosis of spinal disorder other than degenerative disc at the involved level;
* Has a symptomatic disc herniation at more than one lumbar level;
* Requires a herniectomy at more than one lumbar level;
* Has a disc degeneration at the treated and adjacent levels > Grade IV (Pfirrmann, 2001);
* Has a decrease of disc height ≥ 30% as measured by the center of the disc space, and compared to the disc space at the next superior spinal level;
* Has Modic changes on MRI greater than Grade I at the target level;
* Has Modic changes on MRI at the adjacent levels;
* Has an advanced degree of retrolisthesis as shown by lateral X-rays (> 25%, i.e. grade I as per Meyerding);
* Has a clinical evidence of lysis, antero listhesis or scoliosis (Cobb angle more than 10°);
* Has signs of segmental instability: more than 4 mm of translation or more than 10° angular motion between adjacent end plates (comparing flexion and extension views);
* Has congenital or iatrogenic posterior element insufficiency (e.g. facet resection, spondylolysis, pars fracture, or Spinal Bifida Occulta);
* Has had any previous lumbar spine surgery;
* Has a Waddell signs of inorganic behaviour score greater than or equal to 3;
* Has evidence of an active disruptive psychiatric disorder, cognitive impairment or other known condition, significant enough to impact the perception of pain, precludes surgical procedure, clinical evaluation and/or ability to evaluate treatment outcome as determined by investigator;
* Has a known allergy to silicone, polyethylene, or titanium;
* Is an alcohol and /or drug abuser, as defined by currently undergoing treatment for alcohol and/or drug abuse;
* Has obesity defined by BMI greater than or equal to 35;
* Inability to complete the questionnaires;
* Planned pregnancy during the course of the study;
* Previous enrollment into a spine study;
* Vulnerable patients or unable to exercise free informed consent;

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2006-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdiand Krappel, Dr., Principal Investigator — Spitalzentrum Oberwallis, Brig
Locations (19):
- Belgium (4):
  - Cliniques Universitaires Bruxelles Hôpital Erasme, Brussels
  - AZ Sint-Lucas, Ghent
  - Hôpital de la Citadelle, Liège
  - AZ Sint-Elisabeth Hospital, Zottegem
- University Hospital Olomouc, dept of Neurosurgery, Olomouc, Czechia
- Germany (3):
  - Otto-Von-Guericke Universität, Magdeburg
  - CA NCH Klinikum rechts der Isar/München, München
  - Medizinisches Zentrum Kreis Aachen, Würselen
- Italy (2):
  - Anthea Casa di Cura, Bari
  - Istituto Ortopedico Galeazzi, Milan
- St. Luke Hospital, University of Rzeszow, dept of Neurosurgery, Tarnów, Poland
- Spain (2):
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital de León, León
- Switzerland (3):
  - Hôpital Fribourgeois, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Hirslanden Klinik St. Anna, Lucerne
- United Kingdom (3):
  - Chase Farm Hospital, Enfield
  - St. Georges Hospital, London
  - Greater Manchester Neuroscience Center, Salford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 patients were enrolled but not randomized:
  6 were excluded due to eligibility criteria not met, and 1 was excluded due to non-compliance issue.
Period: Overall Study
Arm/Group | Investigational Group | Control Group
Started | 75 (4 pts were removed due to compliance issue. 2 pts were randomized but not treated (non-eligible)) | 71 (5 pts were removed due to compliance issue. 1 pt was randomized but not treated (Non-eligible))
6 Weeks Follow-up | 72 (Withdrawn (n=1). Visit not done (n=2)) | 67 (Withdrawn (n=2). Visit not done (n=2))
3 Months Follow-up | 72 (Visit not done (n=2)) | 68 (Visit not done (n=1))
6 Months Follow-up | 71 (Visit not done (n=3)) | 63 (Withdrawn (n=3). Visit not done (n=3))
12 Months Follow-up | 68 (Withdrawn(n=4). Visit not done (n=2)) | 60 (Withdrawn (n=1). Visit not done (n=4). Lost to follow-up (n=1))
24 Months Follow up | 57 (Withdrawn (n=5) Accidental death (n=1) Lost to follow up (n=7)) | 58 (Withdrawn (n=3). Lost to follow-up (n=3))
Completed | 57 | 58
Not Completed | 18 | 13
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 0 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group | Control Group | Total
Number analyzed (Participants) | 75 | 71 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (10) | 40.7 (10.7) | 41.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate a Statistically Significant Difference in the Relief of Back Pain Between Both Treatment Groups. The Endpoint Will be the Difference Between Baseline and 6-month of the Patient's Back-pain Score on a Visual Analogue Scale (VAS).
Description: The endpoint will be the difference between baseline and 6 months of the patient's back-pain score on a Visual Analogue Scale (VAS). A standardized visual analogue scale (0cm-10cm; with 0cm meaning 'no pain' and 10cm meaning 'worst possible pain') will be used. Large values of the VAS score represent large degree of pain. Large (negative) change in VAS score (6 months - baseline) represents large relief of pain. For treated subjects, all analyses except the safety analyses, Intent-To-Treat population will serve as the primary analysis dataset.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 68 | 63
units on a scale | -3.97 (2.55) | -3.37 (3.15)
Statistical Analysis 1: Comparison: Investigational Group vs Control Group; The null-hypothesis: Ho: Δ VAS DIAM = Δ VAS Control will be tested against the alternative hypothesis:HA: Δ VAS DIAM ≠ Δ VAS Control.Where Δ is the average decrease in VAS score (baseline - 6 months). A minimal sample size of 240 analyzable patients is required to demonstrate with 80% power a difference in back pain reduction that is significant at the 95% level, comparing DIAM and Control groups. 268 patients will be enroll to allow of up to 10% attrition; Test type: Superiority or Other; p = 0.228, t-test, 2 sided; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.59 to 0.38]

2. Secondary Outcome: To Demonstrate a Statistically Significant Difference in the Reduction of Disability Between Both Treatment Groups. The Endpoint Will be the Difference Between Baseline and 12 Months of the Patient's Score on the Oswestry Disability Index (ODI).
Description: The endpoint will be the difference between baseline and 12 months of the patient's score on the Oswestry Disability Index (ODI).
  The ODI is a low back pain disability questionnaire used to measure a patient's permanent functional disability in a scale from 0 to 50 (when all the 10 sections are answered); large ODI scores indicate large disability.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: patient's score
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 68 | 61
patient's score | -38.55 (20.10) | -37.19 (22.61)
Statistical Analysis 1: Comparison: Investigational Group vs Control Group; The null-hypothesis(Ho: Δ ODI DIAM = Δ ODI Control) will be tested against the alternative hypothesis (HA: Δ ODI DIAM ≠ Δ ODI Control). Δ ODI DIAM = average change in the ODI (12 months - baseline) in the DIAM treated patient group and Δ VAS Control =average change in the ODI in the Control group; Test type: Superiority or Other; p = 0.719, t-test, 2 sided; Mean Difference (Net) = -1.36, 95% CI 2-sided [-8.80 to 6.08]

ADVERSE EVENTS:
Time Frame: 2 years
Description: For safety analyses, the "As-Treated" population has been used as the primary analysis dataset. In this analysis, a patient was grouped as investigational group (implanted with a DIAM device) or control group according to the true treatment the patient has received, regardless of randomization.
Arm/Group | Investigational Group | Control Group
Serious Adverse Events (participants affected / at risk) | 15/73 | 19/71
Other Adverse Events (participants affected / at risk) | 44/73 | 40/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=73) | Control Group (N=71)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ACCIDENTAL DEATH (General disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 2 (3)
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=73) | Control Group (N=71)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 (19) | 20 (25)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 18 (18) | 11 (12)
SCIATICA (Nervous system disorders) | 4 (4) | 2 (2)
CARDIAC VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DURAL TEAR (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GASTRIC PH DECREASED (Investigations) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOTONIA (Nervous system disorders) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
PROSTATISM (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The current study was limited by not reaching the target enrollment. Because of the low patient recruitment rate, despite major efforts by the investigators and sponsor, enrollment was stopped prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less